CLINICAL TRIAL: NCT03941262
Title: Phase 1, Open-Label, Safety Study of Escalating Doses of Ex Vivo Expanded, Autologous Natural Killer Cells in Patients With Pathologically Confirmed Cancer Refractory to Conventional Therapy
Brief Title: Safety of SNK01 in Subjects With Pathologically Confirmed Metastatic and/or Unresectable Cancer Refractory to Conventional Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NKGen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNK01-US01
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Refractory Cancer; Metastatic Cancer; Recurrent Cancer; Unresectable Carcinoma; Solid Tumor, Adult; Advanced Cancer; Advanced Solid Tumor
Keywords: Natural killer cell; NK cell; Expanded natural killer cell; Immunotherapy; Cancer; Metastatic cancer; Advanced solid tumor; Refractory cancer; Recurrent cancer; Unresectable carcinoma; Solid tumor; Neoplasms
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Recurrence | interventions — avelumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 - Low dose SNK01 (Experimental): SNK01 (low dose) administered once a week for five weeks.
  Interventions: Biological: SNK01
- Cohort 2 - Medium dose SNK01 (Experimental): SNK01 (medium dose) administered once a week for five weeks.
  Interventions: Biological: SNK01
- Cohort 3 - High dose SNK01 (Experimental): SNK01 (high dose) administered once a week for five weeks.
  Interventions: Biological: SNK01
- Cohort 4 - SNK01 with avelumab (Experimental): SNK01 (high dose) administered in combination with avelumab once every two weeks (14-day cycle) for five cycles.
  Interventions: Biological: SNK01; Drug: Avelumab
- Cohort 4 - SNK01 with pembrolizumab (Experimental): SNK01 (high dose) administered in combination with pembrolizumab once every three weeks (21-day cycle) for five cycles.
  Interventions: Biological: SNK01; Drug: Pembrolizumab

INTERVENTIONS:
Biological: SNK01 — Patient-specific ex vivo expanded autologous natural killer cells
Drug: Avelumab — Avelumab is a humanized monoclonal antibody immune checkpoint blockade immunotherapy that targets the programmed cell death-ligand 1 (PD-L1).
  Other Names: Bavencio
  Arms: Cohort 4 - SNK01 with avelumab
Drug: Pembrolizumab — Pembrolizumab is a humanized monoclonal antibody immune checkpoint blockade immunotherapy that targets the programmed cell death receptor-1 (PD-1).
  Other Names: Keytruda
  Arms: Cohort 4 - SNK01 with pembrolizumab

SUMMARY:
The purpose of the study is to evaluate the safety and preliminary efficacy of SNK01 (autologous natural killer cell), as a single agent and in combination with avelumab or pembrolizumab, for the treatment of subjects with advanced and/or metastatic refractory cancer that has failed three or more prior lines of conventional standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent signed by patient, obtained prior to study enrollment.
* Males and females ages 18 to 75 years, inclusive.
* Pathologically confirmed diagnosis of refractory cancer that has failed three or more prior lines of conventional standard of care therapy.
* Diagnosed with any histologically confirmed malignancy whose disease is confirmed to be metastatic and/or unresectable for which standard curative or beneficial treatments are no longer effective.
* Eastern Cooperative Oncology Group (ECOG) performance status <2.
* At least 4 weeks since any prior systemic therapy (excluding corticosteroid therapy) to treat the underlying malignancy (standard or investigational).
* At least 2 weeks since prior palliative radiotherapy.
* Adequate bone marrow function:

  * Neutrophils: 2.0-8.0 K/uL
  * Platelet Count: 140-440 K/uL
  * Hemoglobin: 10.0-18.0 g/dL
  * No ongoing transfusion requirements
* Adequate hepatic function:

  * Serum total bilirubin < 1.5 x upper limit of normal (ULN)
  * Serum albumin ≥ 3.0 g/dL
  * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN
  * International normalized ratio (INR) ≤ 1.5 x ULN
* Adequate renal function with creatinine ≤ 2.0 mg/dL.
* Negative pregnancy test for women of childbearing potential and use of effective contraception (hormonal or barrier method of birth control) during study.

Exclusion Criteria:

* Pregnant and/or lactating females.
* Life expectancy of less than three months.
* Currently being treated by "biological therapy" as defined by the National Cancer Institute (example: checkpoint inhibitors, adoptive cell transfer, monoclonal antibodies, treatment vaccines, cytokines, Bacillus Calmette-Guerin (BCG), chimeric antigen receptor T cell therapy (CAR-T), and natural killer cell therapy).
* Patients tested positive for hepatitis B and/or C surface antigen.
* High fever or any active or unresolved infection, including human immunodeficiency virus (HIV) positive.
* Autoimmune disease requiring therapy; immunodeficiency, or any disease process requiring immunosuppressive therapy.
* Prior clinical trial requiring patient to receive an investigational drug within two weeks of enrollment.
* Congestive heart failure, unstable angina or other underlying cardiac disease; history of thrombosis currently requiring anticoagulation.
* Mental or psychological illness preventing cooperation with treatment, efficacy evaluations, or unable to understand the informed consent process.
* Subjects who have undergone prior organ transplantation, including allogeneic stem-cell transplantation.
* Adult subjects who lack capacity to consent for themselves and for whom consent must be provided by a legally authorized representative.
* For SNK01+avelumab arm only: Subjects with prior hypersensitivity to avelumab or its excipients, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* For SNK01+avelumab arm only: Subjects with a significant immune-mediated adverse event due to a prior checkpoint inhibitor immunotherapy that led to permanent discontinuation of the therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
To assess the safety profile | Up to 6 months
  Assessed by the incidence and severity of dose limiting toxicity (DLT) and other adverse events graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI-CTCAE), Version 5.0, or the cytokine release syndrome revised grading system.

SECONDARY OUTCOMES:
To assess clinical objective response rate (ORR) of SNK01 in patients with refractory cancer | Up to 12 months
  Objective response rate (ORR) is defined by the percentage of subjects who achieve a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.
To assess clinical objective response rate (ORR) of SNK01 in combination with avelumab in patients with refractory cancer | Up to 12 months
  Objective response rate (ORR) is defined by the percentage of subjects who achieve a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.
To assess clinical objective response rate (ORR) of SNK01 in combination with pembrolizumab in patients with refractory cancer | Up to 12 months
  Objective response rate (ORR) is defined by the percentage of subjects who achieve a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chang, MPH, Study Director — NKGen Biotech, Inc.
Locations (1):
- Sarcoma Oncology Research Center, Santa Monica, California, United States